CLINICAL TRIAL: NCT03070652
Title: What Are the Effects of Supporting Early Parenting by Increasing the Understanding of the Infant? A Randomized Community Based Trial
Brief Title: What Are the Effects of Supporting Early Parenting by Increasing the Understanding of the Infant?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Hanne Kronborg, Associate Professor, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SUN-Aarhus-2017- 653
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Parent-Child Relations
Keywords: attachment; bonding psychological

ARMS (2):
- NBO, Newborn behavioral observation (Experimental): In the intervention group new parents will receive the NBO delivered in connection with the examination of the newborn in a shared observation with the parents in the homevisit of the health visitor 3 weeks post partum
  Interventions: Behavioral: NBO, Newborn behavioral observation
- Practice as usual (Experimental): In the comparison group new parents will receive practice as usual due to the examination of their newborn in the homevisit of the health visitor 3 weeks post partum
  Interventions: Behavioral: Practice as usual

INTERVENTIONS:
Behavioral: NBO, Newborn behavioral observation
  Arms: NBO, Newborn behavioral observation
Behavioral: Practice as usual
  Arms: Practice as usual

SUMMARY:
Key research question This project addresses the following key research question: What are the short and long term effects on child and family outcomes of a universal intervention delivered by a Health Visitor addressing the newborn´s behavior in a shared observation with the parents (NBO)? The aim is to enhance the parent's sensitivity to their infants' unique capacities and thereby create an early parental understanding for the individual infant's strengths as well as its needs.

Hypothesis concerning main outcomes

Universal Health Visiting with facilitation of the early relationship building introduced by the NBO to an intervention group of new families will- when compared to a control group of new families who receive health visitor support as usual:

* Improve sensitive responsive parenting to the infant's behavior, needs for feeding and comfort, and rise understanding of parental influence on the infants' self-regulatory capacities
* Increase parental confidence and reduce experiences of stress and symptoms of depression among new mothers and fathers
* Improve the infant's self-regulatory capacities regarding sleep, crying, feeding and engaging in social interactions, being more cooperative
* Enhance the sensitive early parent/infant relationship
* Improve exclusive breastfeeding duration and delay introduction to solid food

Method The project is formed as a community based randomized trial. The complexity in community based intervention research is the existence of two target groups, in this case: 1) the primary study population of new parents that receive the supportive intervention and 2) the secondary study population of Health Visitors that deliver the supportive intervention. The complication of catching the effects in a universal approach will be addressed through a variety of outcomes that capture both the aspect and the development of the infant, the mother and the father and the interactions.

Recruitment and randomization Four medium-sized municipalities will join in the trial. To avoid side-effects the districts of the Health Visitors in the participating municipalities will be regarded as clusters. A restricted randomization procedure is decided to achieve balance in the two study arms because of a relatively small number of clusters (n=17) with huge differences in birth rate. The criteria for the restricted randomization is a geographical balance with all participating municipalities represented by both intervention and comparison districts and a numerical balance with expected number of births attempted between the intervention and comparison group. An external data manager performed the entire procedure.

Study population The primary study population is formed by new families, mothers and fathers and their infant/s. Substantiated in that we are operating with a community based universal intervention with no side effects and we seek to measure the effect in a natural population we will have no exclusion criteria except parents or infants affiliated to special treatment elsewhere.

In the study population of new parents there will be subgroups: First time parents will represent around 40 %, around 6 % will have given premature birth, 2% twin birth, 10-14% of the mothers and 7-8% of the fathers will suffer from birth depression in the postnatal period, and 7-20% will have a cultural background other than Danish depending on geographical area.

A subgroup of 100 first-time mothers in each group of intervention and comparison are drawn consecutively among responders for video recording in the middle of the project period after specified characteristic criteria with regard to first-time-, depressed- and given premature birth.

Data and data-collection Data will be collected from two sources: (1) self-reported data from the new parents collected via questionnaire; (2) observational data from video recordings, Infant CARE-Index. Questionnaire data will be delivered and collected though an internet based system. Participating mothers and fathers will receive separate questionnaires at 1-2 weeks postpartum (baseline data), 3 months postpartum, 9 months follow-up, 18 months follow-up. Videos are recorded at 3 months post-partum (corrected age for premature infants) with 3 minutes of unstructured time together; (Infant CARE Index). All data will be linked via the Danish Personal Register (CPR) identifier. To minimize bias introduced by data collection, data will be collected in the same way and with the same timing in the intervention and comparison groups.

Data Analysis Intention to treat analysis will be used to detect the effect of the community based intervention where motivation and participation may vary in both the primary and secondary study population. Supplemental analysis will be performed to identify an intervention effect for subgroups and marginal groups of parents according to parity, preterm delivery, and depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

The primary study population is formed by new families, mothers and fathers and their newborn/s. Substantiated in that we are operating with a community based universal intervention with no side effects and we seek to measure the effect in a natural population we will have no exclusion criteria

Exclusion Criteria:

* except parents or infants affiliated to special treatment elsewhere.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2566 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Karitane parenting confidence scale, KPCS. Change is being assessed. | measured at 2 weeks, 3 and 9 months post partum
  Parents´sense of confidence
Infant Care Index | measured 4 months post partum
  Parental sensitivity, responsiveness and early parent infant relationship
Ages & States questionnarie, ASQ-SE. Change is being assessed. | measured at 2 weeks, 3 and 9 months post partum
  Infant's self-regulatory capacities, understanding of parental influence on the infants' self-regulatory capacities

SECONDARY OUTCOMES:
The Major Depression Inventory (MDI10) | measured at 2 weeks, 3 and 9 months post partum
  Depression associated with parenting
Breast-feeding period in weeks | measured at 3 and 9 months
  The duration of full breastfeeding following birth measured in weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Kronborg, Principal Investigator — Section of Nursing, Department of Public Health, Aarhus University
Locations (1):
- Institute of Publich Health, Department of Nursing Science, University of Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Kristensen IH, Juul S, Kronborg H. What are the effects of supporting early parenting by newborn behavioral observations (NBO)? A cluster randomised trial. BMC Psychol. 2020 Oct 16;8(1):107. doi: 10.1186/s40359-020-00467-5. PMID 33076981
- [Derived] Kristensen IH, Kronborg H. What are the effects of supporting early parenting by enhancing parents' understanding of the infant? Study protocol for a cluster-randomized community-based trial of the Newborn Behavioral Observation (NBO) method. BMC Public Health. 2018 Jul 4;18(1):832. doi: 10.1186/s12889-018-5747-4. PMID 29973172